CLINICAL TRIAL: NCT01206062
Title: Systolic Blood Pressure Intervention Trial
Acronym: SPRINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, David Reboussin, Principal Investigator, Coordinating Center, Wake Forest University Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPRINT; 268200900040C-1-0-1 (NIH)
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Hypertension
Keywords: blood pressure; antihypertensive; systolic; diastolic; heart failure; myocardial infarction; stroke; chronic kidney disease; dementia; cognitive decline
MeSH Terms: conditions — Hypertension; Systolic Murmurs; Heart Murmurs; Heart Failure; Myocardial Infarction; Stroke; Renal Insufficiency, Chronic; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Control of SBP (Experimental): Participants randomized into the Intensive BP arm will have a goal of SBP <120 mm Hg. 2-drug therapy initiated in most Intensive participants; age ≥75 years and SBP 130-139 mm Hg on 0-1 drug; may begin with 1 drug, but add second at 1 month if SBP ≥130 mm Hg; drugs added and/or titrated at each visit (monthly) to achieve SBP <120 mm Hg; at periodic "milepost" visits: addition of another drug "required" if not at goal.
  Interventions: Drug: Intensive control of SBP
- Standard Control of SBP (Active Comparator): Participants randomized into the Standard arm will have a goal of SBP <140 mm Hg. Intensify therapy if SBP ≥160 mm Hg @ 1 visit; ≥140 mm Hg @ 2 consecutive visits; Down-titration if SBP <130 mm Hg @ 1 visit; <135 mm Hg @ 2 consecutive visits
  Interventions: Drug: Standard control of SBP

INTERVENTIONS:
Drug: Intensive control of SBP — Participants in the Intensive arm have a goal of SBP <120 mm Hg. Use of once-daily antihypertensive agents will be encouraged unless alternative frequency is indicated/necessary. One or more medications from the following classes of agents will be provided by the study for use in managing participants in both randomization groups to achieve study goals:
  Angiotension converting enzyme (ACE)-inhibitors Angiotension receptor blockers (ARBs) Direct vasodilators Thiazide-type diuretics Loop diuretics Potassium-sparing diuretics Beta-blockers Sustained-release calcium channel blockers (CCBs) Alpha1-receptor blockers Sympatholytics
  Combination products will be available, depending on cost, utility, or donations from pharmaceutical companies.
  Other Names: Lower target for SBP; Comparison of standard SBP control to a target of 120 mm Hg
  Arms: Intensive Control of SBP
Drug: Standard control of SBP — Participants in the Standard BP arm have a goal of SBP <140 mm Hg. The same medications used in the Intensive BP arm will be used for the Standard BP arm.
  Other Names: Control of SBP to a target of 140 mm Hg
  Arms: Standard Control of SBP

SUMMARY:
Elevated blood pressure (BP) is an important public health concern. It is highly prevalent, the prevalence may be increasing, and it is a risk factor for several adverse health outcomes, especially coronary heart disease, stroke, heart failure, chronic kidney disease, and decline in cognitive function. The Systolic Blood Pressure Intervention Trial (SPRINT) is a 2-arm, multicenter, randomized clinical trial designed to test whether a treatment program aimed at reducing systolic blood pressure (SBP) to a lower goal than currently recommended will reduce cardiovascular disease (CVD) risk.

DETAILED DESCRIPTION:
SPRINT strived to enroll about 9250 participants aged ≥ 50 years with SBP ≥130 mm Hg and at least one additional CVD risk factor. The trial compared the effects of randomization to a treatment program of an intensive SBP goal with randomization to a treatment program of a standard goal. Target SBP goals were <120 vs <140 mm Hg, respectively, to create a minimum mean difference of 10 mm Hg between the two randomized groups. The primary hypothesis was that CVD event rates would be lower in the intensive arm. Participants were recruited at approximately 90 clinics within 5 clinical center networks (CCNs) over approximately a 2-year period, and were followed for 4-6 years.

A total of 9361 participants were enrolled. NIH stopped the blood pressure intervention earlier than originally planned in order to quickly disseminate the significant preliminary results. Follow-up for cognitive and kidney outcomes continues during the post-intervention phase through May 2018.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years old

Systolic blood pressure of

* 130 - 180 mm Hg on 0 or 1 medication
* 130 - 170 mm Hg on up to 2 medications
* 130 - 160 mm Hg on up to 3 medications
* 130 - 150 mm Hg on up to 4 medications

Risk (one or more of the following)

1. Presence of clinical or subclinical cardiovascular disease other than stroke
2. CKD, defined as eGFR 20 - 59 ml/min/1.73m2
3. A Framingham Risk Score for 10-year CVD risk ≥ 15%
4. Age greater than 75 years

Exclusion Criteria:

* An indication for a specific BP lowering medication that the person is not taking and the person has not been documented to be intolerant of the medication class.
* Known secondary cause of hypertension that causes concern regarding safety of the protocol.
* One minute standing SBP < 110 mm Hg.
* Proteinuria in the following ranges (based on a measurement within the past 6 months)

  * 24 hour urinary protein excretion ≥1 g/day, or
  * 24 hour urinary albumin excretion ≥ 600 mg/day, or
  * spot urine protein/creatinine ratio ≥ 1 g/g creatinine, or
  * spot urine albumin/creatinine ratio ≥ 600 mg/g creatinine, or
  * urine dipstick ≥ 2+ protein
* Arm circumference too large or small to allow accurate blood pressure measurement with available devices
* Diabetes mellitus,
* History of stroke (not CE or stenting)
* Diagnosis of polycystic kidney disease
* Glomerulonephritis treated with or likely to be treated with immunosuppressive therapy
* eGFR < 20 ml/min /1.73m2 or end-stage renal disease (ESRD)
* Cardiovascular event or procedure (as defined above as clinical CVD for study entry) or hospitalization for unstable angina within last 3 months
* Symptomatic heart failure within the past 6 months or left ventricular ejection fraction (by any method) < 35%
* A medical condition likely to limit survival to less than 3 years or a malignancy other than non-melanoma skin cancer within the last 2 years
* Any factors judged by the clinic team to be likely to limit adherence to interventions.
* Failure to obtain informed consent from participant
* Currently participating in another clinical trial (intervention study). Note: Patient must wait until the completion of his/her activities or the completion of the other trial before being screened for SPRINT.
* Living in the same household as an already randomized SPRINT participant
* Any organ transplant
* Unintentional weight loss > 10% in last 6 months
* Pregnancy, currently trying to become pregnant, or of child-bearing potential and not using birth control.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9361 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Reboussin, PhD, Principal Investigator — Wake Forest University Health Sciences; Jackson T Wright, MD, Principal Investigator — Case Western Reserve University; Alfred Cheung, MD, Principal Investigator — University of Utah; Suzanne Oparil, MD, Principal Investigator — University of Alabama at Birmingham; Mike Rocco, MD, Principal Investigator — Wake Forest University Health Sciences; Bill Cushman, MD, Principal Investigator — Memphis VA Medical Center
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ambrosius WT, Sink KM, Foy CG, Berlowitz DR, Cheung AK, Cushman WC, Fine LJ, Goff DC Jr, Johnson KC, Killeen AA, Lewis CE, Oparil S, Reboussin DM, Rocco MV, Snyder JK, Williamson JD, Wright JT Jr, Whelton PK; SPRINT Study Research Group. The design and rationale of a multicenter clinical trial comparing two strategies for control of systolic blood pressure: the Systolic Blood Pressure Intervention Trial (SPRINT). Clin Trials. 2014 Oct;11(5):532-46. doi: 10.1177/1740774514537404. Epub 2014 Jun 5. PMID 24902920
- [Background] Ramsey TM, Snyder JK, Lovato LC, Roumie CL, Glasser SP, Cosgrove NM, Olney CM, Tang RH, Johnson KC, Still CH, Gren LH, Childs JC, Crago OL, Summerson JH, Walsh SM, Perdue LH, Bankowski DM, Goff DC; SPRINT Study Research Group. Recruitment strategies and challenges in a large intervention trial: Systolic Blood Pressure Intervention Trial. Clin Trials. 2016 Jun;13(3):319-30. doi: 10.1177/1740774516631735. Epub 2016 Feb 24. PMID 26911833
- [Result] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Derived] Wang S, Wang J, Wang Y, Xu X, Gu H, Xie W, Cai L, Zhang J, Wang T, Zhao Z, Li M, Zheng J, Xu M, Lu J, Bi Y, Xu Y. Intensive blood pressure control and risks of cognitive outcomes in patients with new-onset orthostatic hypotension. Age Ageing. 2026 Jan 3;55(1):afag005. doi: 10.1093/ageing/afag005. PMID 41609319
- [Derived] Wang Y, Tang S, Li M, Chen M. Fluctuations in adherence to antihypertensive medication and cardiovascular outcomes: a secondary analysis of the SPRINT trial. Hypertens Res. 2026 Jan 15. doi: 10.1038/s41440-025-02538-9. Online ahead of print. PMID 41540116
- [Derived] Fan C, Wang X, Tao L, Liao Y, Jin L, Shi Q, Wang H, Shi Y, Chang T, Xue Y, Wang J, Yue W, Pan Y, Li Z, Wang Y, Xu M. Insulin Resistance and Blood Pressure Control on Cognitive Outcomes. Hypertension. 2026 Jan;83(1):199-211. doi: 10.1161/HYPERTENSIONAHA.125.24666. Epub 2025 Nov 26. PMID 41293821
- [Derived] Chen WH, Yang C, Chen YT, Li ZJ, Guan K, Li JJ, Huang RC. Systolic Blood Pressure Time in Target Range and Acute Kidney Injury in Patients With Hypertension. Hypertension. 2025 Dec;82(12):2218-2226. doi: 10.1161/HYPERTENSIONAHA.125.25511. Epub 2025 Oct 9. PMID 41064861
- [Derived] Li N, Yang Z, Yuan Q, Cheng W. A Risk Stratification Model for Predicting Benefits of Intensive Blood Pressure Treatment: Analysis of the Systolic Blood Pressure Intervention Trial. J Clin Hypertens (Greenwich). 2025 Aug;27(8):e70098. doi: 10.1111/jch.70098. PMID 40751458
- [Derived] Chen X, Wang L, Jiang Y, Tang W, Xiao J, Deng W, Ren X, Li C. Interplay between triglyceride-glucose index and cardiovascular events in hypertensive patients with controlled blood pressure (SBP<140 mmHg): insights from the SPRINT trial. Front Endocrinol (Lausanne). 2025 Jul 16;16:1508667. doi: 10.3389/fendo.2025.1508667. eCollection 2025. PMID 40741171
- [Derived] Pewowaruk R, Jaeger BC, Hughes TM, Upadhya B, Kitzman DW, Supiano MA, Gepner AD. Effects of Blood Pressure Control on Arterial Stiffness Mechanisms in SPRINT: A Randomized Controlled Trial. Hypertension. 2025 Jun;82(6):1004-1011. doi: 10.1161/HYPERTENSIONAHA.124.24816. Epub 2025 Apr 22. PMID 40260539
- [Derived] Zhang Y, Zheng W, Jiang C, Hao W, Gong W, Yan Y, Wang X, Ma C, Nie S. Sex-Specific Association between Systolic Blood Pressure Time in Target Range and Cardiovascular Outcomes: A Post-Hoc Analysis of the SPRINT Trial. Rev Cardiovasc Med. 2025 Mar 18;26(3):26262. doi: 10.31083/RCM26262. eCollection 2025 Mar. PMID 40160598
- [Derived] Zheng W, Li S, Jiang C, Hao W, Ai H, Wang X, Ma C, Nie S. Effect of Intensive Blood Pressure Control and Comorbidity Status on the Prognosis of Patients With Hypertension: Insights From SPRINT. J Am Heart Assoc. 2025 Mar 18;14(6):e036719. doi: 10.1161/JAHA.124.036719. Epub 2025 Mar 17. PMID 40094181
- [Derived] Reboussin DM, Gaussoin SA, Pajewski NM, Jaeger BC, Sachs B, Rapp SR, Supiano MA, Cleveland ML, Hunter V, Demons JL, Ogrocki PK, Lerner AJ, Chelune GJ, Wadley VG, Scales ML, Woolard NF, Perdue LH, Callahan KE, Williamson JD. Long-Term Effect of Intensive vs Standard Blood Pressure Control on Mild Cognitive Impairment and Probable Dementia in SPRINT. Neurology. 2025 Feb 11;104(3):e213334. doi: 10.1212/WNL.0000000000213334. Epub 2025 Jan 16. PMID 39819096
- [Derived] Sible IJ, Nation DA. Comparison of visit-to-visit blood pressure variability and time in target range in predicting risk for cognitive outcomes in the SPRINT trial. J Alzheimers Dis. 2025 Jan;103(2):396-405. doi: 10.1177/13872877241303378. Epub 2024 Dec 16. PMID 39686614
- [Derived] Li M, Zhao S, Yu S, Maimaitiaili R, Xu Y, Li Y, Zhao Y, Zhang Y. Association Between Systolic Blood Pressure Time in Target Range Indices and Adverse Cardiovascular Outcomes. JACC Adv. 2024 Oct 18;3(11):101350. doi: 10.1016/j.jacadv.2024.101350. eCollection 2024 Nov. PMID 39497947
- [Derived] Kazibwe R, Ahmad MI, Singh S, Chen LY, Soliman EZ. Effect of Intensive Blood Pressure Lowering on the Risk of Incident Silent Myocardial Infarction: A Post Hoc Analysis of a Randomized Controlled Trial. Ann Noninvasive Electrocardiol. 2024 Nov;29(6):e70018. doi: 10.1111/anec.70018. PMID 39359164
- [Derived] Pajewski NM, Beddhu S, Bress AP, Chang TI, Chertow GM, Cheung AK, Cushman WC, Freedman BI, Greene T, Johnson KC, Jaeger BC, Tamura MK, Lewis CE, Rahman M, Reboussin DM, Rocco MV, Williamson JD, Whelton PK, Wright JT Jr, Drawz PE, Ix JH. The Legacy Effect of Intensive versus Standard BP Control on the Incidence of Needing Dialysis or Kidney Transplantation. J Am Soc Nephrol. 2024 Dec 1;35(12):1737-1745. doi: 10.1681/ASN.0000000000000459. Epub 2024 Jul 30. PMID 39078712
- [Derived] Liu X, Lin B, Yao S, Pan Z. Impact of Anemia on Cardiovascular Events and All-Cause Death Among Participants Who Received Intense Blood Pressure Treatment: A Secondary Analysis of SPRINT. Rev Cardiovasc Med. 2024 Jan 8;25(1):6. doi: 10.31083/j.rcm2501006. eCollection 2024 Jan. PMID 39077655
- [Derived] Zhang Z, Li L, Zhang Z, Hu Z, Xiong Y, Zhou L, Yao Y. Electrocardiographic tracking of left ventricular hypertrophy in hypertension: incidence and prognostic outcomes from the SPRINT trial. Clin Hypertens. 2024 Jul 1;30(1):17. doi: 10.1186/s40885-024-00275-8. PMID 38946010
- [Derived] Mirzai S, Persits I, Kazibwe R, Gabani M, Seals A, Singleton MJ, Rikhi R, Chevli PA, Carbone S, Tang WHW, Yeboah J, Williamson JD, Kitzman DW, Herrington DM, Shapiro MD. Relationship Between Sarcopenia and Intensive Blood Pressure Control Efficacy and Safety: A Secondary Analysis of SPRINT. Hypertension. 2024 Aug;81(8):e77-e87. doi: 10.1161/HYPERTENSIONAHA.124.23011. Epub 2024 Jun 17. PMID 38881460
- [Derived] Kazibwe R, Schaich CL, Muhammad AI, Epiu I, Namutebi JH, Chevli PA, Kazibwe J, Hughes T, Rikhi RR, Shapiro MD, Yeboah J. Effect of vigorous-intensity physical activity on incident cognitive impairment in high-risk hypertension. Alzheimers Dement. 2024 Jul;20(7):4602-4612. doi: 10.1002/alz.13887. Epub 2024 Jun 6. PMID 38842100
- [Derived] Wang Z, Li W, Jiang C, Wang J, Hua C, Tang Y, Zhang H, Liu X, Wang Y, Gao M, Lv Q, Dong J, Ma C, Du X. Association between blood pressure variability and risk of kidney function decline in hypertensive patients without chronic kidney disease: a post hoc analysis of Systolic Blood Pressure Intervention Trial study. J Hypertens. 2024 Jul 1;42(7):1203-1211. doi: 10.1097/HJH.0000000000003715. Epub 2024 Mar 8. PMID 38690929
- [Derived] Sible IJ, Nation DA. Blood Pressure Variability and Plasma Alzheimer's Disease Biomarkers in the SPRINT Trial. J Alzheimers Dis. 2024;97(4):1851-1860. doi: 10.3233/JAD-230930. PMID 38306042
- [Derived] Li W, Wang Z, Jiang C, Hua C, Tang Y, Zhang H, Liu X, Zheng S, Wang Y, Gao M, Lv Q, Dong J, Ma C, Du X. Effect of Intensive Blood Pressure Control on Cardiovascular Outcomes in Cancer Survivors. Hypertension. 2024 Mar;81(3):620-628. doi: 10.1161/HYPERTENSIONAHA.123.22194. Epub 2024 Jan 2. PMID 38164752
- [Derived] Jia X, Nambi V, Berry JD, Dalmacy D, Ascher SB, Taylor AA, Hoogeveen RC, de Lemos JA, Ballantyne CM. High-Sensitivity Cardiac Troponins I and T and Cardiovascular Outcomes: Findings from the Systolic Blood Pressure Intervention Trial (SPRINT). Clin Chem. 2024 Feb 7;70(2):414-424. doi: 10.1093/clinchem/hvad209. PMID 38084941
- [Derived] Huang X, Deng S, Xie W, Zheng F. Time in target range of systolic blood pressure and cognitive outcomes in patients with hypertension. J Am Geriatr Soc. 2024 Feb;72(2):423-432. doi: 10.1111/jgs.18641. Epub 2023 Nov 2. PMID 37916517
- [Derived] Kern KC, Nasrallah IM, Bryan RN, Reboussin DM, Wright CB. Intensive systolic blood pressure treatment remodels brain perivascular spaces: A secondary analysis of the Systolic Pressure Intervention Trial (SPRINT). Neuroimage Clin. 2023;40:103513. doi: 10.1016/j.nicl.2023.103513. Epub 2023 Sep 23. PMID 37774646
- [Derived] King JB, Berchie RO, Derington CG, Marcum ZA, Scharfstein DO, Greene TH, Herrick JS, Jacobs JA, Zheutlin AR, Bress AP, Cohen JB. New Users of Angiotensin II Receptor Blocker-Versus Angiotensin-Converting Enzyme Inhibitor-Based Antihypertensive Medication Regimens and Cardiovascular Disease Events: A Secondary Analysis of ACCORD-BP and SPRINT. J Am Heart Assoc. 2023 Sep 5;12(17):e030311. doi: 10.1161/JAHA.123.030311. Epub 2023 Aug 30. PMID 37646208
- [Derived] Wang J, Jiang C, Li S, Wang Z, Wang Y, Lai Y, Wang Z, Lv W, Bai Y, Yang Z, Guo Q, Huang L, He L, Guo X, Li S, Liu N, Jiang C, Tang R, Long D, Du X, Sang C, Dong J, Ma C. Systolic Blood Pressure Time in Target Range and Incident Atrial Fibrillation in Patients With Hypertension: Insights From the SPRINT Trial. Hypertension. 2023 Nov;80(11):2306-2314. doi: 10.1161/HYPERTENSIONAHA.123.21651. Epub 2023 Aug 17. PMID 37589154
- [Derived] de Havenon A, Smith EE, Sharma R, Falcone GJ, Bangad A, Prabhakaran S, Sheth KN. Improvement in the Prediction of Cerebrovascular Events With White Matter Hyperintensity. J Am Heart Assoc. 2023 Jul 4;12(13):e029374. doi: 10.1161/JAHA.123.029374. Epub 2023 Jun 22. PMID 37345754
- [Derived] Sible IJ, Nation DA. Blood Pressure Variability and Cerebral Perfusion Decline: A Post Hoc Analysis of the SPRINT MIND Trial. J Am Heart Assoc. 2023 Jun 20;12(12):e029797. doi: 10.1161/JAHA.123.029797. Epub 2023 Jun 10. PMID 37301768
- [Derived] King JB, Derington CG, Herrick JS, Jacobs JA, Zheutlin AR, Conroy MB, Cushman WC, Bress AP. Single-Pill Combination Product Availability of the Antihypertensive Regimens Used for Intensive Systolic Blood Pressure Treatment in the Systolic Blood Pressure Intervention Trial. Hypertension. 2023 Aug;80(8):1749-1758. doi: 10.1161/HYPERTENSIONAHA.123.21132. Epub 2023 Jun 8. PMID 37288570
- [Derived] Ghazi L, Shen J, Ying J, Derington CG, Cohen JB, Marcum ZA, Herrick JS, King JB, Cheung AK, Williamson JD, Pajewski NM, Bryan N, Supiano M, Sonnen J, Weintraub WS, Greene TH, Bress AP. Identifying Patients for Intensive Blood Pressure Treatment Based on Cognitive Benefit: A Secondary Analysis of the SPRINT Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2314443. doi: 10.1001/jamanetworkopen.2023.14443. PMID 37204788
- [Derived] Li S, Jiang C, Wang Y, Lai Y, Zhao M, Li Q, Bai Y, Dai W, Guo Q, He L, Guo X, Wang W, Li S, Liu N, Jiang C, Tang R, Sang C, Long D, Du X, Dong J, Anderson CS, Ma C. Systolic Blood Pressure Time in Target Range and Cognitive Outcomes: Insights From the SPRINT MIND Trial. Hypertension. 2023 Aug;80(8):1628-1636. doi: 10.1161/HYPERTENSIONAHA.122.20711. Epub 2023 May 11. PMID 37165869
- [Derived] Frimodt-Moller EK, Vittinghoff E, Kaur G, Biering-Sorensen T, Soliman EZ, Marcus GM. Association Between Intensive vs Standard Blood Pressure Control and Incident Left Ventricular Conduction Disease: A Post Hoc Analysis of the SPRINT Randomized Clinical Trial. JAMA Cardiol. 2023 Jun 1;8(6):612-616. doi: 10.1001/jamacardio.2023.0845. PMID 37133829
- [Derived] Wang Z, Wang Q, Pei J, Wang X, Li Y, Yan J, Du X. Association Between the Frailty and Cognitive Impairment Among Patients With Hypertension-A Post Hoc Analysis of the SPRINT Trial. J Am Heart Assoc. 2023 Apr 4;12(7):e028736. doi: 10.1161/JAHA.122.028736. Epub 2023 Mar 28. PMID 36974773
- [Derived] Lin B, Liu X, Yao S, Pan Z. Intensive Blood Pressure Control and Diabetes Mellitus Incidence for Patients with Impaired Fasting Glucose: A Secondary Analysis of SPRINT. Int J Hypertens. 2023 Mar 16;2023:7533353. doi: 10.1155/2023/7533353. eCollection 2023. PMID 36968629
- [Derived] Kern KC, Nasrallah IM, Bryan RN, Reboussin DM, Wright CB. Intensive Systolic Blood Pressure Treatment Remodels Brain Perivascular Spaces: A Secondary Analysis of SPRINT. medRxiv [Preprint]. 2023 Feb 23:2023.02.22.23286329. doi: 10.1101/2023.02.22.23286329. PMID 36865252
- [Derived] Rashid T, Li K, Toledo JB, Nasrallah I, Pajewski NM, Dolui S, Detre J, Wolk DA, Liu H, Heckbert SR, Bryan RN, Williamson J, Davatzikos C, Seshadri S, Launer LJ, Habes M. Association of Intensive vs Standard Blood Pressure Control With Regional Changes in Cerebral Small Vessel Disease Biomarkers: Post Hoc Secondary Analysis of the SPRINT MIND Randomized Clinical Trial. JAMA Netw Open. 2023 Mar 1;6(3):e231055. doi: 10.1001/jamanetworkopen.2023.1055. PMID 36857053
- [Derived] Jiang C, Li S, Wang Y, Lai Y, Bai Y, Zhao M, He L, Kong Y, Guo X, Li S, Liu N, Jiang C, Tang R, Sang C, Long D, Du X, Dong J, Anderson CS, Ma C. Diastolic Blood Pressure and Intensive Blood Pressure Control on Cognitive Outcomes: Insights From the SPRINT MIND Trial. Hypertension. 2023 Mar;80(3):580-589. doi: 10.1161/HYPERTENSIONAHA.122.20112. Epub 2023 Jan 23. PMID 36688305
- [Derived] Sheng CS, Wang D, Yuan J, Cheng Y, Sun S, Yang Y, Miao Y, Wang W, Tian J, Bloomgarden ZT. CVD risk in non-albuminuric chronic kidney disease in hypertensive, non-diabetic subjects: A post-hoc analysis from SPRINT. Front Cardiovasc Med. 2022 Dec 7;9:977938. doi: 10.3389/fcvm.2022.977938. eCollection 2022. PMID 36568559
- [Derived] Derington CG, Bress AP, Moran AE, Weintraub WS, Herrick JS, Cushman WC, Kronish IM, Stults B, Shimbo D, Muntner P, Greene T, Bates JT, Chang TI, Katz LA, Rehman SU, Roumie CL, Tamariz L, King JB. Antihypertensive Medication Regimens Used in the Systolic Blood Pressure Intervention Trial. Hypertension. 2023 Mar;80(3):590-597. doi: 10.1161/HYPERTENSIONAHA.122.20373. Epub 2022 Dec 15. PMID 36519451
- [Derived] Sible IJ, Nation DA. Blood Pressure Variability and Cognitive Decline: A Post Hoc Analysis of the SPRINT MIND Trial. Am J Hypertens. 2023 Feb 24;36(3):168-175. doi: 10.1093/ajh/hpac128. PMID 36448621
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Jaeger BC, Bress AP, Bundy JD, Cheung AK, Cushman WC, Drawz PE, Johnson KC, Lewis CE, Oparil S, Rocco MV, Rapp SR, Supiano MA, Whelton PK, Williamson JD, Wright JT Jr, Reboussin DM, Pajewski NM. Longer-Term All-Cause and Cardiovascular Mortality With Intensive Blood Pressure Control: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2022 Nov 1;7(11):1138-1146. doi: 10.1001/jamacardio.2022.3345. PMID 36223105
- [Derived] Kim DH, Tatsuoka C, Chen Z, Wright JT Jr, Odden MC, Beddhu S, Bellows BK, Bress A, Carson T, Cushman WC, Johnson KC, Morisky DE, Punzi H, Tamariz L, Yang S, Wei LJ. Intensive Versus Standard Blood Pressure Lowering and Days Free of Cardiovascular Events and Serious Adverse Events: a Post Hoc Analysis of Systolic Blood Pressure Intervention Trial. J Gen Intern Med. 2022 Nov;37(15):3797-3804. doi: 10.1007/s11606-022-07753-5. Epub 2022 Aug 9. PMID 35945470
- [Derived] Cushman WC, Ringer RJ, Rodriguez CJ, Evans GW, Bates JT, Cutler JA, Hawfield A, Kitzman DW, Nasrallah IM, Oparil S, Nord J, Papademetriou V, Servilla K, Van Buren P, Whelton PK, Whittle J, Wright JT Jr; SPRINT Research Group. Blood Pressure Intervention and Control in SPRINT. Hypertension. 2022 Sep;79(9):2071-2080. doi: 10.1161/HYPERTENSIONAHA.121.17233. Epub 2022 Jun 29. PMID 35766041
- [Derived] Jiang C, Lai Y, Du X, Wang Y, Li S, He L, Hu R, Lv Q, Wu J, Feng L, Ning M, Ruan Y, Li X, Jia C, Dai W, Guo X, Jiang C, Tang R, Sang C, Long D, Arima H, Dong J, Anderson CS, Ma C. Effects of intensive blood pressure control on cardiovascular and cognitive outcomes in patients with atrial fibrillation: insights from the SPRINT trial. Europace. 2022 Oct 13;24(10):1560-1568. doi: 10.1093/europace/euac059. PMID 35640916
- [Derived] Inoue K, Watson KE, Kondo N, Horwich T, Hsu W, Bui AAT, Duru OK. Association of Intensive Blood Pressure Control and Living Arrangement on Cardiovascular Outcomes by Race: Post Hoc Analysis of SPRINT Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e222037. doi: 10.1001/jamanetworkopen.2022.2037. PMID 35285922
- [Derived] Dolui S, Detre JA, Gaussoin SA, Herrick JS, Wang DJJ, Tamura MK, Cho ME, Haley WE, Launer LJ, Punzi HA, Rastogi A, Still CH, Weiner DE, Wright JT Jr, Williamson JD, Wright CB, Bryan RN, Bress AP, Pajewski NM, Nasrallah IM. Association of Intensive vs Standard Blood Pressure Control With Cerebral Blood Flow: Secondary Analysis of the SPRINT MIND Randomized Clinical Trial. JAMA Neurol. 2022 Apr 1;79(4):380-389. doi: 10.1001/jamaneurol.2022.0074. PMID 35254390
- [Derived] Parcha V, Heindl B, Kalra R, Bress A, Rao S, Pandey A, Gower B, Irvin MR, McDonald MN, Li P, Arora G, Arora P. Genetic European Ancestry and Incident Diabetes in Black Individuals: Insights From the SPRINT Trial. Circ Genom Precis Med. 2022 Feb;15(1):e003468. doi: 10.1161/CIRCGEN.121.003468. Epub 2022 Jan 28. PMID 35089798
- [Derived] Zheutlin AR, Mondesir FL, Derington CG, King JB, Zhang C, Cohen JB, Berlowitz DR, Anstey DE, Cushman WC, Greene TH, Ogedegbe O, Bress AP. Analysis of Therapeutic Inertia and Race and Ethnicity in the Systolic Blood Pressure Intervention Trial: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2143001. doi: 10.1001/jamanetworkopen.2021.43001. PMID 35006243
- [Derived] de Vries TI, Stam-Slob MC, Peters RJG, van der Graaf Y, Westerink J, Visseren FLJ. Impact of a Patient's Baseline Risk on the Relative Benefit and Harm of a Preventive Treatment Strategy: Applying Trial Results in Clinical Decision Making. J Am Heart Assoc. 2022 Jan 4;11(1):e017605. doi: 10.1161/JAHA.120.017605. Epub 2021 Dec 22. PMID 34935407
- [Derived] Pareek M, Vaduganathan M, Byrne C, Mikkelsen AD, Kristensen AMD, Biering-Sorensen T, Kragholm KH, Omar M, Olsen MH, Bhatt DL. Intensive blood pressure control in patients with a history of heart failure: the Systolic Blood Pressure Intervention Trial (SPRINT). Eur Heart J Cardiovasc Pharmacother. 2022 May 5;8(3):E12-E14. doi: 10.1093/ehjcvp/pvab085. No abstract available. PMID 34902012
- [Derived] Upadhya B, Willard JJ, Lovato LC, Rocco MV, Lewis CE, Oparil S, Cushman WC, Bates JT, Bello NA, Aurigemma G, Johnson KC, Rodriguez CJ, Raj DS, Rastogi A, Tamariz L, Wiggers A, Kitzman DW; SPRINT Research Group. Incidence and Outcomes of Acute Heart Failure With Preserved Versus Reduced Ejection Fraction in SPRINT. Circ Heart Fail. 2021 Dec;14(12):e008322. doi: 10.1161/CIRCHEARTFAILURE.121.008322. Epub 2021 Nov 26. PMID 34823375
- [Derived] Pajewski NM, Elahi FM, Tamura MK, Hinman JD, Nasrallah IM, Ix JH, Miller LM, Launer LJ, Wright CB, Supiano MA, Lerner AJ, Sudduth TL, Killeen AA, Cheung AK, Reboussin DM, Wilcock DM, Williamson JD. Plasma amyloid beta, neurofilament light chain, and total tau in the Systolic Blood Pressure Intervention Trial (SPRINT). Alzheimers Dement. 2022 Aug;18(8):1472-1483. doi: 10.1002/alz.12496. Epub 2021 Nov 17. PMID 34786815
- [Derived] Byrne C, Pareek M, Vaduganathan M, Biering-Sorensen T, Krogager ML, Kragholm KH, Steensig K, Mortensen MB, Mishra SR, McCullough MJ, Desai NR, Torp-Pedersen C, Olsen MH, Bhatt DL. Serum Potassium and Mortality in High-Risk Patients: SPRINT. Hypertension. 2021 Nov;78(5):1586-1594. doi: 10.1161/HYPERTENSIONAHA.121.17736. Epub 2021 Oct 4. PMID 34601970
- [Derived] Kurella Tamura M, Gaussoin S, Pajewski NM, Zaharchuk G, Freedman BI, Rapp SR, Auchus AP, Haley WE, Oparil S, Kendrick J, Roumie CL, Beddhu S, Cheung AK, Williamson JD, Detre JA, Dolui S, Bryan RN, Nasrallah IM; SPRINT Research Group. Kidney Disease, Hypertension Treatment, and Cerebral Perfusion and Structure. Am J Kidney Dis. 2022 May;79(5):677-687.e1. doi: 10.1053/j.ajkd.2021.07.024. Epub 2021 Sep 17. PMID 34543687
- [Derived] Berry JD, Nambi V, Ambrosius WT, Chen H, Killeen AA, Taylor A, Toto RD, Soliman EZ, McEvoy JW, Pandey A, Joshi PH, Blankenberg S, Kitzman DW, Ballantyne CM, de Lemos JA. Associations of High-Sensitivity Troponin and Natriuretic Peptide Levels With Outcomes After Intensive Blood Pressure Lowering: Findings From the SPRINT Randomized Clinical Trial. JAMA Cardiol. 2021 Dec 1;6(12):1397-1405. doi: 10.1001/jamacardio.2021.3187. PMID 34468696
- [Derived] Cheng Y, Li J, Ren X, Wang D, Yang Y, Miao Y, Sheng CS, Tian J. Visit-to-visit office blood pressure variability combined with Framingham risk score to predict all-cause mortality: A post hoc analysis of the systolic blood pressure intervention trial. J Clin Hypertens (Greenwich). 2021 Aug;23(8):1516-1525. doi: 10.1111/jch.14314. Epub 2021 Jul 3. PMID 34216524
- [Derived] Alborzi A, Attar A, Sayadi M, Nouri F. The Effects of Intensive Blood Pressure Control on Cardiovascular Outcomes Based on 10-Year ASCVD Risk Score: An Analysis of a Clinical Trial. Cardiol Res Pract. 2021 May 11;2021:6635345. doi: 10.1155/2021/6635345. eCollection 2021. PMID 34055403
- [Derived] SPRINT Research Group; Lewis CE, Fine LJ, Beddhu S, Cheung AK, Cushman WC, Cutler JA, Evans GW, Johnson KC, Kitzman DW, Oparil S, Rahman M, Reboussin DM, Rocco MV, Sink KM, Snyder JK, Whelton PK, Williamson JD, Wright JT Jr, Ambrosius WT. Final Report of a Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2021 May 20;384(20):1921-1930. doi: 10.1056/NEJMoa1901281. PMID 34010531
- [Derived] Bellows BK, Zhang Y, Zhang Z, Lloyd-Jones DM, Bress AP, King JB, Kolm P, Cushman WC, Johnson KC, Tamariz L, Oelsner EC, Shea S, Newman AB, Ives DG, Couper D, Moran AE, Weintraub WS. Estimating Systolic Blood Pressure Intervention Trial Participant Posttrial Survival Using Pooled Epidemiologic Cohort Data. J Am Heart Assoc. 2021 May 18;10(10):e020361. doi: 10.1161/JAHA.120.020361. Epub 2021 May 6. PMID 33955229
- [Derived] Bress AP, Greene T, Derington CG, Shen J, Xu Y, Zhang Y, Ying J, Bellows BK, Cushman WC, Whelton PK, Pajewski NM, Reboussin D, Beddu S, Hess R, Herrick JS, Zhang Z, Kolm P, Yeh RW, Basu S, Weintraub WS, Moran AE; SPRINT Research Group. Patient Selection for Intensive Blood Pressure Management Based on Benefit and Adverse Events. J Am Coll Cardiol. 2021 Apr 27;77(16):1977-1990. doi: 10.1016/j.jacc.2021.02.058. PMID 33888247
- [Derived] Wang X, Pei J, Zheng K, Hu X. High-density lipoprotein cholesterol levels are associated with major adverse cardiovascular events in male but not female patients with hypertension. Clin Cardiol. 2021 May;44(5):723-730. doi: 10.1002/clc.23606. Epub 2021 Mar 30. PMID 33786851
- [Derived] Upadhya B, Pajewski NM, Rocco MV, Hundley WG, Aurigemma G, Hamilton CA, Bates JT, He J, Chen J, Chonchol M, Glasser SP, Hung AM, Pisoni R, Punzi H, Supiano MA, Toto R, Taylor A, Kitzman DW; SPRINT Research Group. Effect of Intensive Blood Pressure Control on Aortic Stiffness in the SPRINT-HEART. Hypertension. 2021 May 5;77(5):1571-1580. doi: 10.1161/HYPERTENSIONAHA.120.16676. Epub 2021 Mar 29. PMID 33775127
- [Derived] Nasrallah IM, Gaussoin SA, Pomponio R, Dolui S, Erus G, Wright CB, Launer LJ, Detre JA, Wolk DA, Davatzikos C, Williamson JD, Pajewski NM, Bryan RN; SPRINT Research Group. Association of Intensive vs Standard Blood Pressure Control With Magnetic Resonance Imaging Biomarkers of Alzheimer Disease: Secondary Analysis of the SPRINT MIND Randomized Trial. JAMA Neurol. 2021 May 1;78(5):568-577. doi: 10.1001/jamaneurol.2021.0178. PMID 33683313
- [Derived] Vaduganathan M, Pareek M, Kristensen AMD, Biering-Sorensen T, Byrne C, Almarzooq Z, Olesen TB, Olsen MH, Bhatt DL. Prevention of heart failure events with intensive versus standard blood pressure lowering across the spectrum of kidney function and albuminuria: a SPRINT substudy. Eur J Heart Fail. 2021 Mar;23(3):384-392. doi: 10.1002/ejhf.1971. Epub 2020 Aug 20. PMID 33448580
- [Derived] Shah C, Srinivasan D, Erus G, Schmitt JE, Agarwal A, Cho ME, Lerner AJ, Haley WE, Kurella Tamura M, Davatzikos C, Bryan RN, Fan Y, Nasrallah IM. Changes in brain functional connectivity and cognition related to white matter lesion burden in hypertensive patients from SPRINT. Neuroradiology. 2021 Jun;63(6):913-924. doi: 10.1007/s00234-020-02614-6. Epub 2021 Jan 6. PMID 33404789
- [Derived] Xu X, Meng X, Oka SI. Long-Term Habitual Vigorous Physical Activity Is Associated With Lower Visit-to-Visit Systolic Blood Pressure Variability: Insights From the SPRINT Trial. Am J Hypertens. 2021 May 22;34(5):463-466. doi: 10.1093/ajh/hpaa198. PMID 33245323
- [Derived] Rocco MV, Comeau ME, Marion MC, Freedman BI, Hawfield AT, Langefeld CD; SPRINT Research Group*. Effects of Intensive Systolic Blood Pressure Control on All-Cause Hospitalizations. Hypertension. 2020 Dec;76(6):1717-1724. doi: 10.1161/HYPERTENSIONAHA.120.15868. Epub 2020 Oct 26. PMID 33100049
- [Derived] Rapp SR, Gaussoin SA, Sachs BC, Chelune G, Supiano MA, Lerner AJ, Wadley VG, Wilson VM, Fine LJ, Whittle JC, Auchus AP, Beddhu S, Berlowitz DR, Bress AP, Johnson KC, Krousel-Wood M, Martindale-Adams J, Miller EC, Rifkin DE, Snyder JK, Tamariz L, Wolfgram DF, Cleveland ML, Yang M, Nichols LO, Bryan RN, Reboussin DM, Williamson JD, Pajewski NM; SPRINT Research Group. Effects of intensive versus standard blood pressure control on domain-specific cognitive function: a substudy of the SPRINT randomised controlled trial. Lancet Neurol. 2020 Nov;19(11):899-907. doi: 10.1016/S1474-4422(20)30319-7. PMID 33098800
- [Derived] Drawz PE, Agarwal A, Dwyer JP, Horwitz E, Lash J, Lenoir K, McWilliams A, Oparil S, Rahbari-Oskoui F, Rahman M, Parkulo MA, Pemu P, Raj DS, Rocco M, Soman S, Thomas G, Tuot DS, Whelton PK, Pajewski NM. Concordance Between Blood Pressure in the Systolic Blood Pressure Intervention Trial and in Routine Clinical Practice. JAMA Intern Med. 2020 Dec 1;180(12):1655-1663. doi: 10.1001/jamainternmed.2020.5028. PMID 33044494
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623
- [Derived] Frary JMC, Pareek M, Byrne C, Vaduganathan M, Biering-Sorensen T, Rujic D, Kragholm KH, Olesen TB, Olsen MH, Bhatt DL. Intensive blood pressure control appears to be effective and safe in patients with peripheral artery disease: the Systolic Blood Pressure Intervention Trial. Eur Heart J Cardiovasc Pharmacother. 2021 May 23;7(3):e38-e40. doi: 10.1093/ehjcvp/pvaa102. No abstract available. PMID 32853332
- [Derived] Borazjani R, Kojuri J, Abdi-Ardekani A, Izadpanah P, Dehghani P, Sayadi M, Attar A. Pharmacological treatment of high-normal blood pressure (prehypertension) in high-risk patients for primary prevention of cardiovascular events. J Clin Hypertens (Greenwich). 2020 Sep;22(9):1627-1634. doi: 10.1111/jch.13994. Epub 2020 Aug 20. PMID 32815661
- [Derived] Krogager ML, Pareek M, Kragholm KH, Byrne C, Vaduganathan M, Biering-Sorensen T, Rujic D, Olesen TB, Olsen MH, Bhatt DL. Intensive vs. standard blood pressure control and vascular procedures: insights from the Systolic Blood Pressure Intervention Trial (SPRINT). Eur Heart J Cardiovasc Pharmacother. 2021 May 23;7(3):e35-e37. doi: 10.1093/ehjcvp/pvaa093. No abstract available. PMID 32722801
- [Derived] Parcha V, Patel N, Kalra R, Kim J, Gutierrez OM, Arora G, Arora P. Incidence and Implications of Atrial Fibrillation/Flutter in Hypertension: Insights From the SPRINT Trial. Hypertension. 2020 Jun;75(6):1483-1490. doi: 10.1161/HYPERTENSIONAHA.120.14690. Epub 2020 May 4. PMID 32362231
- [Derived] Soliman EZ, Rahman AF, Zhang ZM, Rodriguez CJ, Chang TI, Bates JT, Ghazi L, Blackshear JL, Chonchol M, Fine LJ, Ambrosius WT, Lewis CE. Effect of Intensive Blood Pressure Lowering on the Risk of Atrial Fibrillation. Hypertension. 2020 Jun;75(6):1491-1496. doi: 10.1161/HYPERTENSIONAHA.120.14766. Epub 2020 May 4. PMID 32362229
- [Derived] Collard D, Brouwer TF, Olde Engberink RHG, Zwinderman AH, Vogt L, van den Born BH. Initial Estimated Glomerular Filtration Rate Decline and Long-Term Renal Function During Intensive Antihypertensive Therapy: A Post Hoc Analysis of the SPRINT and ACCORD-BP Randomized Controlled Trials. Hypertension. 2020 May;75(5):1205-1212. doi: 10.1161/HYPERTENSIONAHA.119.14659. Epub 2020 Mar 30. PMID 32223381
- [Derived] Dobre M, Pajewski NM, Beddhu S, Chonchol M, Hostetter TH, Li P, Rahman M, Servilla K, Weiner DE, Wright JT, Raphael KL; SPRINT Research Group. Serum bicarbonate and cardiovascular events in hypertensive adults: results from the Systolic Blood Pressure Intervention Trial. Nephrol Dial Transplant. 2020 Aug 1;35(8):1377-1384. doi: 10.1093/ndt/gfz149. PMID 32163578
- [Derived] Vaduganathan M, Claggett BL, Juraschek SP, Solomon SD. Assessment of Long-term Benefit of Intensive Blood Pressure Control on Residual Life Span: Secondary Analysis of the Systolic Blood Pressure Intervention Trial (SPRINT). JAMA Cardiol. 2020 May 1;5(5):576-581. doi: 10.1001/jamacardio.2019.6192. PMID 32101262
- [Derived] Juraschek SP, Taylor AA, Wright JT Jr, Evans GW, Miller ER 3rd, Plante TB, Cushman WC, Gure TR, Haley WE, Moinuddin I, Nord J, Oparil S, Pedley C, Roumie CL, Whittle J, Wiggers A, Finucane C, Anne Kenny R, Appel LJ, Townsend RR; SPRINT Research Group. Orthostatic Hypotension, Cardiovascular Outcomes, and Adverse Events: Results From SPRINT. Hypertension. 2020 Mar;75(3):660-667. doi: 10.1161/HYPERTENSIONAHA.119.14309. Epub 2020 Jan 27. PMID 31983312
- [Derived] Roumie CL, Hung AM, Russell GB, Basile J, Kreider KE, Nord J, Ramsey TM, Rastogi A, Sweeney ME, Tamariz L, Kostis WJ, Williams JS, Zias A, Cushman WC; SPRINT Research Group. Blood Pressure Control and the Association With Diabetes Mellitus Incidence: Results From SPRINT Randomized Trial. Hypertension. 2020 Feb;75(2):331-338. doi: 10.1161/HYPERTENSIONAHA.118.12572. Epub 2019 Dec 23. PMID 31865790
- [Derived] Pajewski NM, Berlowitz DR, Bress AP, Callahan KE, Cheung AK, Fine LJ, Gaussoin SA, Johnson KC, King J, Kitzman DW, Kostis JB, Lerner AJ, Lewis CE, Oparil S, Rahman M, Reboussin DM, Rocco MV, Snyder JK, Still C, Supiano MA, Wadley VG, Whelton PK, Wright JT Jr,, Williamson JD. Intensive vs Standard Blood Pressure Control in Adults 80 Years or Older: A Secondary Analysis of the Systolic Blood Pressure Intervention Trial. J Am Geriatr Soc. 2020 Mar;68(3):496-504. doi: 10.1111/jgs.16272. Epub 2019 Dec 16. PMID 31840813
- [Derived] Upadhya B, Lovato LC, Rocco M, Lewis CE, Oparil S, Cushman WC, Kostis JB, Rodriguez CJ, Cho ME, Cloud LW, Rastogi A, Rosendorff C, Kitzman DW; SPRINT Research Group. Heart Failure Prevention in Older Patients Using Intensive Blood Pressure Reduction: Potential Role of Diuretics. JACC Heart Fail. 2019 Dec;7(12):1032-1041. doi: 10.1016/j.jchf.2019.08.018. PMID 31779925
- [Derived] Berlowitz DR, Foy C, Conroy M, Evans GW, Olney CM, Pisoni R, Powell JR, Gure TR, Shorr RI. Impact of Intensive Blood Pressure Therapy on Concern about Falling: Longitudinal Results from the Systolic Blood Pressure Intervention Trial (SPRINT). J Am Geriatr Soc. 2020 Mar;68(3):614-618. doi: 10.1111/jgs.16264. Epub 2019 Nov 28. PMID 31778222
- [Derived] Lee CL, Wang JS. Systolic blood pressure trajectory and cardiovascular outcomes: An analysis using data in the Systolic Blood Pressure Intervention Trial. Int J Clin Pract. 2020 Mar;74(3):e13450. doi: 10.1111/ijcp.13450. Epub 2019 Dec 6. PMID 31755625
- [Derived] Leitao L, Soares-Dos-Reis R, Neves JS, Baptista RB, Bigotte Vieira M, Mc Causland FR. Intensive Blood Pressure Treatment Reduced Stroke Risk in Patients With Albuminuria in the SPRINT Trial. Stroke. 2019 Dec;50(12):3639-3642. doi: 10.1161/STROKEAHA.119.026316. Epub 2019 Oct 22. PMID 31637971
- [Derived] Sundstrom J, Karmali KN. The case for absolute cardiovascular risk-based blood pressure-lowering treatment decisions: data from the SPRINT trial. J Hum Hypertens. 2020 Jul;34(7):544-545. doi: 10.1038/s41371-019-0260-5. Epub 2019 Sep 23. No abstract available. PMID 31548621
- [Derived] Byrne C, Pareek M, Vaduganathan M, Biering-Sorensen T, Qamar A, Pandey A, Olesen TB, Olsen MH, Bhatt DL. Intensive blood pressure lowering in different age categories: insights from the Systolic Blood Pressure Intervention Trial. Eur Heart J Cardiovasc Pharmacother. 2020 Nov 1;6(6):356-363. doi: 10.1093/ehjcvp/pvz050. PMID 31529024
- [Derived] SPRINT MIND Investigators for the SPRINT Research Group; Nasrallah IM, Pajewski NM, Auchus AP, Chelune G, Cheung AK, Cleveland ML, Coker LH, Crowe MG, Cushman WC, Cutler JA, Davatzikos C, Desiderio L, Doshi J, Erus G, Fine LJ, Gaussoin SA, Harris D, Johnson KC, Kimmel PL, Kurella Tamura M, Launer LJ, Lerner AJ, Lewis CE, Martindale-Adams J, Moy CS, Nichols LO, Oparil S, Ogrocki PK, Rahman M, Rapp SR, Reboussin DM, Rocco MV, Sachs BC, Sink KM, Still CH, Supiano MA, Snyder JK, Wadley VG, Walker J, Weiner DE, Whelton PK, Wilson VM, Woolard N, Wright JT Jr, Wright CB, Williamson JD, Bryan RN. Association of Intensive vs Standard Blood Pressure Control With Cerebral White Matter Lesions. JAMA. 2019 Aug 13;322(6):524-534. doi: 10.1001/jama.2019.10551. PMID 31408137
- [Derived] Lee AK, Katz R, Jotwani V, Garimella PS, Ambrosius WT, Cheung AK, Gren LH, Neyra JA, Punzi H, Raphael KL, Shlipak MG, Ix JH. Distinct Dimensions of Kidney Health and Risk of Cardiovascular Disease, Heart Failure, and Mortality. Hypertension. 2019 Oct;74(4):872-879. doi: 10.1161/HYPERTENSIONAHA.119.13339. Epub 2019 Aug 5. PMID 31378102
- [Derived] Rathi N, Whelton PK, Chertow GM, Cushman WC, Cheung AK, Wei G, Boucher R, Kimmel PL, Bress AP, Kramer HJ, Al-Marji C, Greene T, Beddhu S. Influence of Prediabetes on the Effects of Intensive Systolic Blood Pressure Control on Kidney Events. Am J Hypertens. 2019 Nov 15;32(12):1170-1177. doi: 10.1093/ajh/hpz105. PMID 31257407
- [Derived] Derington CG, Gums TH, Bress AP, Herrick JS, Greene TH, Moran AE, Weintraub WS, Kronish IM, Morisky DE, Trinkley KE, Saseen JJ, Reynolds K, Bates JT, Berlowitz DR, Chang TI, Chonchol M, Cushman WC, Foy CG, Herring CT, Katz LA, Krousel-Wood M, Pajewski NM, Tamariz L, King JB; SPRINT Research Group. Association of Total Medication Burden With Intensive and Standard Blood Pressure Control and Clinical Outcomes: A Secondary Analysis of SPRINT. Hypertension. 2019 Aug;74(2):267-275. doi: 10.1161/HYPERTENSIONAHA.119.12907. Epub 2019 Jul 1. PMID 31256717
- [Derived] Smith SM, Gurka MJ, Winterstein AG, Pepine CJ, Cooper-DeHoff RM. Incidence, prevalence, and predictors of treatment-resistant hypertension with intensive blood pressure lowering. J Clin Hypertens (Greenwich). 2019 Jun;21(6):825-834. doi: 10.1111/jch.13550. Epub 2019 May 7. PMID 31066177
- [Derived] Duan T, Rajpurkar P, Laird D, Ng AY, Basu S. Clinical Value of Predicting Individual Treatment Effects for Intensive Blood Pressure Therapy. Circ Cardiovasc Qual Outcomes. 2019 Mar;12(3):e005010. doi: 10.1161/CIRCOUTCOMES.118.005010. PMID 30857410
- [Derived] Sobieraj P, Lewandowski J, Sinski M, Symonides B, Gaciong Z. Low Diastolic Blood Pressure is Not Related to Risk of First Episode of Stroke in a High-Risk Population: A Secondary Analysis of SPRINT. J Am Heart Assoc. 2019 Feb 19;8(4):e010811. doi: 10.1161/JAHA.118.010811. PMID 30744452
- [Derived] SPRINT MIND Investigators for the SPRINT Research Group; Williamson JD, Pajewski NM, Auchus AP, Bryan RN, Chelune G, Cheung AK, Cleveland ML, Coker LH, Crowe MG, Cushman WC, Cutler JA, Davatzikos C, Desiderio L, Erus G, Fine LJ, Gaussoin SA, Harris D, Hsieh MK, Johnson KC, Kimmel PL, Tamura MK, Launer LJ, Lerner AJ, Lewis CE, Martindale-Adams J, Moy CS, Nasrallah IM, Nichols LO, Oparil S, Ogrocki PK, Rahman M, Rapp SR, Reboussin DM, Rocco MV, Sachs BC, Sink KM, Still CH, Supiano MA, Snyder JK, Wadley VG, Walker J, Weiner DE, Whelton PK, Wilson VM, Woolard N, Wright JT Jr, Wright CB. Effect of Intensive vs Standard Blood Pressure Control on Probable Dementia: A Randomized Clinical Trial. JAMA. 2019 Feb 12;321(6):553-561. doi: 10.1001/jama.2018.21442. PMID 30688979
- [Derived] Rueda-Ochoa OL, Rojas LZ, Ahmad S, van Duijn CM, Ikram MA, Deckers JW, Franco OH, Rizopoulos D, Kavousi M. Impact of cumulative SBP and serious adverse events on efficacy of intensive blood pressure treatment: a randomized clinical trial. J Hypertens. 2019 May;37(5):1058-1069. doi: 10.1097/HJH.0000000000002001. PMID 30444838
- [Derived] Supiano MA, Lovato L, Ambrosius WT, Bates J, Beddhu S, Drawz P, Dwyer JP, Hamburg NM, Kitzman D, Lash J, Lustigova E, Miracle CM, Oparil S, Raj DS, Weiner DE, Taylor A, Vita JA, Yunis R, Chertow GM, Chonchol M. Pulse wave velocity and central aortic pressure in systolic blood pressure intervention trial participants. PLoS One. 2018 Sep 26;13(9):e0203305. doi: 10.1371/journal.pone.0203305. eCollection 2018. PMID 30256784
- [Derived] Beddhu S, Greene T, Boucher R, Cushman WC, Wei G, Stoddard G, Ix JH, Chonchol M, Kramer H, Cheung AK, Kimmel PL, Whelton PK, Chertow GM. Intensive systolic blood pressure control and incident chronic kidney disease in people with and without diabetes mellitus: secondary analyses of two randomised controlled trials. Lancet Diabetes Endocrinol. 2018 Jul;6(7):555-563. doi: 10.1016/S2213-8587(18)30099-8. Epub 2018 Apr 21. PMID 29685860
- [Derived] Dobre M, Gaussoin SA, Bates JT, Chonchol MB, Cohen DL, Hostetter TH, Raphael KL, Taylor AA, Lerner AJ, Wright JT Jr, Rahman M; SPRINT Research Group. Serum Bicarbonate Concentration and Cognitive Function in Hypertensive Adults. Clin J Am Soc Nephrol. 2018 Apr 6;13(4):596-603. doi: 10.2215/CJN.07050717. Epub 2018 Mar 22. PMID 29567858
- [Derived] Johnson KC, Whelton PK, Cushman WC, Cutler JA, Evans GW, Snyder JK, Ambrosius WT, Beddhu S, Cheung AK, Fine LJ, Lewis CE, Rahman M, Reboussin DM, Rocco MV, Oparil S, Wright JT Jr; SPRINT Research Group. Blood Pressure Measurement in SPRINT (Systolic Blood Pressure Intervention Trial). Hypertension. 2018 May;71(5):848-857. doi: 10.1161/HYPERTENSIONAHA.117.10479. Epub 2018 Mar 12. PMID 29531173
- [Derived] Foy CG, Lovato LC, Vitolins MZ, Bates JT, Campbell R, Cushman WC, Glasser SP, Gillespie A, Kostis WJ, Krousel-Wood M, Muhlestein JB, Oparil S, Osei K, Pisoni R, Segal MS, Wiggers A, Johnson KC; SPRINT Study Research Group. Gender, blood pressure, and cardiovascular and renal outcomes in adults with hypertension from the Systolic Blood Pressure Intervention Trial. J Hypertens. 2018 Apr;36(4):904-915. doi: 10.1097/HJH.0000000000001619. PMID 29493562
- [Derived] Vaduganathan M, Pareek M, Qamar A, Pandey A, Olsen MH, Bhatt DL. Baseline Blood Pressure, the 2017 ACC/AHA High Blood Pressure Guidelines, and Long-Term Cardiovascular Risk in SPRINT. Am J Med. 2018 Aug;131(8):956-960. doi: 10.1016/j.amjmed.2017.12.049. Epub 2018 Feb 5. PMID 29421687
- [Derived] Juraschek SP, Miller ER 3rd, Appel LJ. Orthostatic Hypotension and Symptoms in the AASK Trial. Am J Hypertens. 2018 May 7;31(6):665-671. doi: 10.1093/ajh/hpy010. PMID 29370333
- [Derived] Brouwer TF, Vehmeijer JT, Kalkman DN, Berger WR, van den Born BH, Peters RJ, Knops RE. Intensive Blood Pressure Lowering in Patients With and Patients Without Type 2 Diabetes: A Pooled Analysis From Two Randomized Trials. Diabetes Care. 2018 Jun;41(6):1142-1148. doi: 10.2337/dc17-1722. Epub 2017 Dec 6. PMID 29212825
- [Derived] Rocco MV, Sink KM, Lovato LC, Wolfgram DF, Wiegmann TB, Wall BM, Umanath K, Rahbari-Oskoui F, Porter AC, Pisoni R, Lewis CE, Lewis JB, Lash JP, Katz LA, Hawfield AT, Haley WE, Freedman BI, Dwyer JP, Drawz PE, Dobre M, Cheung AK, Campbell RC, Bhatt U, Beddhu S, Kimmel PL, Reboussin DM, Chertow GM; SPRINT Research Group. Effects of Intensive Blood Pressure Treatment on Acute Kidney Injury Events in the Systolic Blood Pressure Intervention Trial (SPRINT). Am J Kidney Dis. 2018 Mar;71(3):352-361. doi: 10.1053/j.ajkd.2017.08.021. Epub 2017 Nov 20. PMID 29162340
- [Derived] Obi Y, Kalantar-Zadeh K, Shintani A, Kovesdy CP, Hamano T. Estimated glomerular filtration rate and the risk-benefit profile of intensive blood pressure control amongst nondiabetic patients: a post hoc analysis of a randomized clinical trial. J Intern Med. 2018 Mar;283(3):314-327. doi: 10.1111/joim.12701. Epub 2017 Nov 19. PMID 29044764
- [Derived] Beddhu S, Chertow GM, Cheung AK, Cushman WC, Rahman M, Greene T, Wei G, Campbell RC, Conroy M, Freedman BI, Haley W, Horwitz E, Kitzman D, Lash J, Papademetriou V, Pisoni R, Riessen E, Rosendorff C, Watnick SG, Whittle J, Whelton PK; SPRINT Research Group. Influence of Baseline Diastolic Blood Pressure on Effects of Intensive Compared With Standard Blood Pressure Control. Circulation. 2018 Jan 9;137(2):134-143. doi: 10.1161/CIRCULATIONAHA.117.030848. Epub 2017 Oct 11. PMID 29021322
- [Derived] Still CH, Rodriguez CJ, Wright JT Jr, Craven TE, Bress AP, Chertow GM, Whelton PK, Whittle JC, Freedman BI, Johnson KC, Foy CG, He J, Kostis JB, Lash JP, Pedley CF, Pisoni R, Powell JR, Wall BM; SPRINT Writing Group. Clinical Outcomes by Race and Ethnicity in the Systolic Blood Pressure Intervention Trial (SPRINT): A Randomized Clinical Trial. Am J Hypertens. 2017 Dec 8;31(1):97-107. doi: 10.1093/ajh/hpx138. PMID 28985268
- [Derived] Kalkman DN, Brouwer TF, Vehmeijer JT, Berger WR, Knops RE, de Winter RJ, Peters RJ, van den Born BH. J Curve in Patients Randomly Assigned to Different Systolic Blood Pressure Targets: An Experimental Approach to an Observational Paradigm. Circulation. 2017 Dec 5;136(23):2220-2229. doi: 10.1161/CIRCULATIONAHA.117.030342. Epub 2017 Sep 22. PMID 28939617
- [Derived] Beddhu S, Rocco MV, Toto R, Craven TE, Greene T, Bhatt U, Cheung AK, Cohen D, Freedman BI, Hawfield AT, Killeen AA, Kimmel PL, Lash J, Papademetriou V, Rahman M, Rastogi A, Servilla K, Townsend RR, Wall B, Whelton PK; SPRINT Research Group. Effects of Intensive Systolic Blood Pressure Control on Kidney and Cardiovascular Outcomes in Persons Without Kidney Disease: A Secondary Analysis of a Randomized Trial. Ann Intern Med. 2017 Sep 19;167(6):375-383. doi: 10.7326/M16-2966. Epub 2017 Sep 5. PMID 28869987
- [Derived] Berlowitz DR, Foy CG, Kazis LE, Bolin LP, Conroy MB, Fitzpatrick P, Gure TR, Kimmel PL, Kirchner K, Morisky DE, Newman J, Olney C, Oparil S, Pajewski NM, Powell J, Ramsey T, Simmons DL, Snyder J, Supiano MA, Weiner DE, Whittle J; SPRINT Research Group. Effect of Intensive Blood-Pressure Treatment on Patient-Reported Outcomes. N Engl J Med. 2017 Aug 24;377(8):733-744. doi: 10.1056/NEJMoa1611179. PMID 28834483
- [Derived] Bress AP, Bellows BK, King JB, Hess R, Beddhu S, Zhang Z, Berlowitz DR, Conroy MB, Fine L, Oparil S, Morisky DE, Kazis LE, Ruiz-Negron N, Powell J, Tamariz L, Whittle J, Wright JT Jr, Supiano MA, Cheung AK, Weintraub WS, Moran AE; SPRINT Research Group. Cost-Effectiveness of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2017 Aug 24;377(8):745-755. doi: 10.1056/NEJMsa1616035. PMID 28834469
- [Derived] Chang TI, Reboussin DM, Chertow GM, Cheung AK, Cushman WC, Kostis WJ, Parati G, Raj D, Riessen E, Shapiro B, Stergiou GS, Townsend RR, Tsioufis K, Whelton PK, Whittle J, Wright JT, Papademetriou V; SPRINT Research Group*. Visit-to-Visit Office Blood Pressure Variability and Cardiovascular Outcomes in SPRINT (Systolic Blood Pressure Intervention Trial). Hypertension. 2017 Oct;70(4):751-758. doi: 10.1161/HYPERTENSIONAHA.117.09788. Epub 2017 Jul 31. PMID 28760939
- [Derived] Soliman EZ, Ambrosius WT, Cushman WC, Zhang ZM, Bates JT, Neyra JA, Carson TY, Tamariz L, Ghazi L, Cho ME, Shapiro BP, He J, Fine LJ, Lewis CE; SPRINT Research Study Group. Effect of Intensive Blood Pressure Lowering on Left Ventricular Hypertrophy in Patients With Hypertension: SPRINT (Systolic Blood Pressure Intervention Trial). Circulation. 2017 Aug 1;136(5):440-450. doi: 10.1161/CIRCULATIONAHA.117.028441. Epub 2017 May 16. PMID 28512184
- [Derived] Patel KK, Arnold SV, Chan PS, Tang Y, Pokharel Y, Jones PG, Spertus JA. Personalizing the Intensity of Blood Pressure Control: Modeling the Heterogeneity of Risks and Benefits From SPRINT (Systolic Blood Pressure Intervention Trial). Circ Cardiovasc Qual Outcomes. 2017 Apr;10(4):e003624. doi: 10.1161/CIRCOUTCOMES.117.003624. PMID 28373269
- [Derived] Upadhya B, Rocco M, Lewis CE, Oparil S, Lovato LC, Cushman WC, Bates JT, Bello NA, Aurigemma G, Fine LJ, Johnson KC, Rodriguez CJ, Raj DS, Rastogi A, Tamariz L, Wiggers A, Kitzman DW; SPRINT Research Group. Effect of Intensive Blood Pressure Treatment on Heart Failure Events in the Systolic Blood Pressure Reduction Intervention Trial. Circ Heart Fail. 2017 Apr;10(4):e003613. doi: 10.1161/CIRCHEARTFAILURE.116.003613. PMID 28364091
- [Derived] Odden MC, Peralta CA, Berlowitz DR, Johnson KC, Whittle J, Kitzman DW, Beddhu S, Nord JW, Papademetriou V, Williamson JD, Pajewski NM; Systolic Blood Pressure Intervention Trial (SPRINT) Research Group. Effect of Intensive Blood Pressure Control on Gait Speed and Mobility Limitation in Adults 75 Years or Older: A Randomized Clinical Trial. JAMA Intern Med. 2017 Apr 1;177(4):500-507. doi: 10.1001/jamainternmed.2016.9104. PMID 28166324
- [Derived] Supiano MA, Williamson JD. Applying the Systolic Blood Pressure Intervention Trial Results to Older Adults. J Am Geriatr Soc. 2017 Jan;65(1):16-21. doi: 10.1111/jgs.14681. Epub 2016 Nov 7. PMID 28111758
- [Derived] Foy CG, Newman JC, Berlowitz DR, Russell LP, Kimmel PL, Wadley VG, Thomas HN, Lerner AJ, Riley WT; SPRINT Study Research Group. Blood Pressure, Sexual Activity, and Dysfunction in Women With Hypertension: Baseline Findings From the Systolic Blood Pressure Intervention Trial (SPRINT). J Sex Med. 2016 Sep;13(9):1333-1346. doi: 10.1016/j.jsxm.2016.06.014. PMID 27555505
- [Derived] Rocco MV, Chapman A, Chertow GM, Cohen D, Chen J, Cutler JA, Diamond MJ, Freedman BI, Hawfield A, Judd E, Killeen AA, Kirchner K, Lewis CE, Pajewski NM, Wall BM, Yee J; SPRINT Research Group. Chronic Kidney Disease Classification in Systolic Blood Pressure Intervention Trial: Comparison Using Modification of Diet in Renal Disease and CKD-Epidemiology Collaboration Definitions. Am J Nephrol. 2016;44(2):130-40. doi: 10.1159/000448722. Epub 2016 Aug 12. PMID 27513312
- [Derived] Williamson JD, Supiano MA, Applegate WB, Berlowitz DR, Campbell RC, Chertow GM, Fine LJ, Haley WE, Hawfield AT, Ix JH, Kitzman DW, Kostis JB, Krousel-Wood MA, Launer LJ, Oparil S, Rodriguez CJ, Roumie CL, Shorr RI, Sink KM, Wadley VG, Whelton PK, Whittle J, Woolard NF, Wright JT Jr, Pajewski NM; SPRINT Research Group. Intensive vs Standard Blood Pressure Control and Cardiovascular Disease Outcomes in Adults Aged >/=75 Years: A Randomized Clinical Trial. JAMA. 2016 Jun 28;315(24):2673-82. doi: 10.1001/jama.2016.7050. PMID 27195814
- [Derived] Thomas HN, Evans GW, Berlowitz DR, Chertow GM, Conroy MB, Foy CG, Glasser SP, Lewis CE, Riley WT, Russell L, Williams O, Hess R; SPRINT Study Group. Antihypertensive medications and sexual function in women: baseline data from the SBP intervention trial (SPRINT). J Hypertens. 2016 Jun;34(6):1224-31. doi: 10.1097/HJH.0000000000000911. PMID 27032074
- [Derived] Tamura MK, Pajewski NM, Bryan RN, Weiner DE, Diamond M, Van Buren P, Taylor A, Beddhu S, Rosendorff C, Jahanian H, Zaharchuk G; SPRINT Study Research Group. Chronic kidney disease, cerebral blood flow, and white matter volume in hypertensive adults. Neurology. 2016 Mar 29;86(13):1208-16. doi: 10.1212/WNL.0000000000002527. Epub 2016 Feb 26. PMID 26920359
- [Derived] Chang TI, Evans G, Cheung AK, Cushman WC, Diamond MJ, Dwyer JP, Huan Y, Kitzman D, Kostis JB, Oparil S, Rastogi A, Roumie CL, Sahay R, Stafford RS, Taylor AA, Wright JT Jr, Chertow GM; SPRINT Study Research Group. Patterns and Correlates of Baseline Thiazide-Type Diuretic Prescription in the Systolic Blood Pressure Intervention Trial. Hypertension. 2016 Mar;67(3):550-5. doi: 10.1161/HYPERTENSIONAHA.115.06851. Epub 2016 Jan 25. PMID 26865200
- [Derived] Cushman WC, Whelton PK, Fine LJ, Wright JT Jr, Reboussin DM, Johnson KC, Oparil S; SPRINT Study Research Group. SPRINT Trial Results: Latest News in Hypertension Management. Hypertension. 2016 Feb;67(2):263-5. doi: 10.1161/HYPERTENSIONAHA.115.06722. Epub 2015 Nov 9. No abstract available. PMID 26553234
- [Derived] Verdecchia P, Angeli F, Reboldi G. The SPRINT trial. J Am Soc Hypertens. 2015 Oct;9(10):750-753. doi: 10.1016/j.jash.2015.09.001. Epub 2015 Sep 9. No abstract available. PMID 26506129

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Control of SBP: Participants randomized into the Intensive BP arm had a goal of SBP <120 mm Hg. 2-drug therapy initiated in most participants; age ≥75 years and SBP 130-139 mm Hg on 0-1 drug; may begin with 1 drug, but add second at 1 month if SBP ≥130 mm Hg; drugs added and/or titrated at each visit (monthly) to achieve SBP <120 mm Hg; at periodic visits: addition of another drug "required" if not at goal.
  Intensive control of SBP: Use of once-daily antihypertensive agents was encouraged unless alternative frequency was necessary. One or more medications from the following classes of agents were provided by the study for use in managing participants in both groups to achieve study goals:
  Angiotension converting enzyme (ACE)-inhibitors Angiotension receptor blockers (ARBs) Direct vasodilators Thiazide-type diuretics Loop diuretics Potassium-sparing diuretics Beta-blockers Sustained-release calcium channel blockers (CCBs) Alpha1-receptor blockers Sympatholytics
- Standard Control of SBP: Participants randomized into the Standard arm had a goal of SBP <140 mm Hg. Intensify therapy if SBP ≥160 mm Hg @ 1 visit; ≥140 mm Hg @ 2 consecutive visits; Down-titration if SBP <130 mm Hg @ 1 visit; <135 mm Hg @ 2 consecutive visits
  Standard control of SBP: The same medications used in the Intensive BP arm will be used for the Standard BP arm.
Period: Overall Study
Arm/Group | Intensive Control of SBP | Standard Control of SBP
Started | 4678 | 4683
Completed | 4678 | 4683
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Control of SBP | Standard Control of SBP | Total
Number analyzed (Participants) | 4678 | 4683 | 9361
Age, Continuous [Mean (Standard Deviation); unit: year]
  Age overall | 67.9 (9.4) | 67.9 (9.5) | 67.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1684 | 1648 | 3332
  Male | 2994 | 3035 | 6029
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race and ethnic group were self-reported.
  Participants
    Non-Hispanic black | 1379 | 1423 | 2802
    Hispanic | 503 | 481 | 984
    Non-Hispanic white | 2698 | 2701 | 5399
    Other | 98 | 78 | 176
Estimated GFR [Mean (Standard Deviation); unit: ml/min/1.73 m2]
  Among all participants | 71.8 (20.7) | 71.7 (20.5) | 71.7 (20.6)
  Among those with estimated GFR >= 60 ml/min/1.73 m | 81.3 (15.5) | 81.1 (15.5) | 81.2 (15.5)
  Among those with estimated GFR < 60 ml/min/1.73 m | 47.8 (9.5) | 47.9 (9.5) | 47.8 (9.5)
Criterion for increased cardiovascular risk [Count of Participants; unit: Participants] — Increased cardiovascular risk was one of the inclusion criteria.
  Chronic kidney disease was defined as an estimated glomerular filtration rate of less than 60 ml per minute per 1.73 m squared of body-surface area.
  Participants
    Age > 75 years | 1317 | 1319 | 2636
    Chronic kidney disease | 1330 | 1316 | 2646
    Cardiovascular disease | 940 | 937 | 1877
    Cardiovascular disease clinical | 779 | 783 | 1562
    Cardiovascular disease subclinical | 247 | 246 | 493
    Framingham CVD risk score >= 15% | 2870 | 2867 | 5737
Black race [Count of Participants; unit: Participants] — Black race includes Hispanic black and black as part of a multiracial identification.
  Participants | 1454 | 1493 | 2947
Baseline BP mm Hg [Mean (Standard Deviation); unit: mm Hg]
  Systolic | 139.7 (15.8) | 139.7 (15.4) | 139.7 (15.6)
  Diastolic | 78.2 (11.9) | 78.0 (12.0) | 78.1 (11.9)
Distribution of systolic blood pressure [Count of Participants; unit: Participants]
  < 132 mm Hg | 1583 | 1553 | 3136
  > 132 mm Hg to < 145 mm Hg | 1489 | 1549 | 3038
  > 145 mm Hg | 1606 | 1581 | 3187
Serum creatinine [Mean (Standard Deviation); unit: mg/dl] | 1.07 (0.34) | 1.08 (0.34) | 1.07 (0.34)
Ratio of urinary albumin (mg) to creatinine (g) [Mean (Standard Deviation); unit: ratio] | 44.1 (178.7) | 41.1 (152.9) | 42.6 (166.3)
Fasting total cholesterol - mg/dl [Mean (Standard Deviation); unit: mg/dl] | 190.2 (41.4) | 190.0 (40.9) | 190.1 (41.2)
Fasting HDL cholesterol - mg/dl [Mean (Standard Deviation); unit: mg/dl] | 52.9 (14.3) | 52.8 (14.6) | 52.9 (14.5)
Fasting total triglycerides - mg/dl [Mean (Standard Deviation); unit: mg/dl] | 124.8 (85.8) | 127.1 (95.0) | 125.9 (90.5)
Fasting plasma glucose - mg/dl [Mean (Standard Deviation); unit: mg/dl] | 98.8 (13.7) | 98.8 (13.4) | 98.8 (13.5)
Statin use [Count of Participants; unit: Participants]
  Statin Use | 1978 | 2076 | 4054
  No Statin Use | 2667 | 2564 | 5231
  Unknown Statin Use | 33 | 43 | 76
Aspirin use [Count of Participants; unit: Participants]
  Aspirin Use | 2406 | 2350 | 4756
  No Aspirin Use | 2255 | 2316 | 4571
  Unknown Aspirin Use | 17 | 17 | 34
Smoking status - no. (%) [Count of Participants; unit: Participants]
  Never smoked | 2050 | 2072 | 4122
  Former smoker | 1977 | 1996 | 3973
  Current smoker | 639 | 601 | 1240
  Missing data | 12 | 14 | 26
Framingham 10-yr cardiovascular disease risk score [Mean (Standard Deviation); unit: probability] — The Framingham Risk Score is a gender-specific algorithm used to estimate the 10-year cardiovascular risk of an individual. It presents risk as the probability of developing coronary heart disease (CHD) within the next 10 years. Individuals with low risk have 10% or less CHD risk at 10 years, with intermediate risk 10-20%, and with high risk 20% or more.
  probability | 24.8 (12.6) | 24.8 (12.5) | 24.8 (12.5)
Body-mass index [Mean (Standard Deviation); unit: kg/m^2] — The body-mass index is the weight in kilograms divided by the square of the height in meters.
  kg/m^2 | 29.9 (5.8) | 29.8 (5.7) | 29.9 (5.8)
Antihypertensive agents - no./patient [Mean (Standard Deviation); unit: agents per patient] | 1.8 (1.0) | 1.8 (1.0) | 1.8 (1.0)
Not using antihypertensive agents - no. (%) [Count of Participants; unit: Participants] | 432 | 450 | 882

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of a Myocardial Infarction (MI), Acute Coronary Syndrome (ACS), Stroke, Heart Failure (HF), or CVD Death
Time Frame: 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Control of SBP | Standard Control of SBP
Number analyzed (Participants) | 4678 | 4683
Participants | 243 | 319
Statistical Analysis 1: Comparison: Intensive Control of SBP vs Standard Control of SBP; Test type: Superiority or Other; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.64 to 0.89]

2. Secondary Outcome: Number of Participants With All-cause Mortality
Time Frame: 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Control of SBP | Standard Control of SBP
Number analyzed (Participants) | 4678 | 4683
Participants | 155 | 210
Statistical Analysis 1: Comparison: Intensive Control of SBP vs Standard Control of SBP; Test type: Superiority or Other; p = 0.003, Regression, Cox; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.60 to 0.90]

3. Secondary Outcome: Number of CKD Participants Who Experienced a 50% Decline From Baseline eGFR
Time Frame: 6 years
Population: Participants with CKD at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Control of SBP | Standard Control of SBP
Number analyzed (Participants) | 1330 | 1316
Participants | 10 | 12
Statistical Analysis 1: Comparison: Intensive Control of SBP vs Standard Control of SBP; Test type: Superiority or Other; p = 0.58, Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.34 to 1.83]

4. Secondary Outcome: Participants Who Developed End Stage Renal Disease
Time Frame: 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Control of SBP | Standard Control of SBP
Number analyzed (Participants) | 4678 | 4683
Participants | 12 | 8

5. Secondary Outcome: Number of Patients With All-cause Dementia
Description: A 3-step process was used ascertain incident cases of all-cause dementia. First, to identify possible cases of dementia a brief Cognition Screening Battery was administered to all participants. Participants who score below the pre-designated screening cut-point for possible cognitive impairment during follow-up were administered a more comprehensive and detailed neurocognitive test battery (the Extended Cognitive Assessment Battery) plus the Functional Assessment Questionnaire (FAQ) which assesses impairments in daily living skills as a result of cognitive impairments. Last, all the above available tests and questionnaire data were submitted to a centralized, web-based system for adjudication by a panel of dementia experts who assigned final study classifications of probable dementia (PD), mild cognitive impairment (MCI) or no impairment (NI).
Time Frame: 6 years
Population: Participants who completed at least 1 cognitive assessment during follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Control of SBP | Standard Control of SBP
Number analyzed (Participants) | 4278 | 4285
Participants | 149 | 176
Statistical Analysis 1: Comparison: Intensive Control of SBP vs Standard Control of SBP; Test type: Superiority or Other; p = .10, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.67 to 1.04]

6. Secondary Outcome: Small Vessel Cerebral Ischemic Disease
Description: Change over 4 years in total white matter lesion volume from baseline Change over 4 years in total brain volume from baseline
  Because of the skewed distribution for WML volume, we first applied an inverse hyperbolic sine transformation (asinh), which is similar to a log transformation but can accommodate values of zero. Linear mixed models, including random effects for participant and MRI facility, were used to estimate the change in WML volume and TBV between the treatment groups, including time since randomization (in days) and intracranial volume as covariates. Because the inverse hyperbolic sine transformation is nonlinear, and given the context of a mixed-effects model, back-transformation to the original scale of cm3 is difficult
Time Frame: 4 years
Population: Of the 670 participants with WML volume measurement at baseline, 462 completed the follow-up MRI. Image quality control requirements were not met for 13 participants with a follow-up MRI scan, resulting in a sample of 449 adults.
Measure: Mean (95% Confidence Interval); unit: asinh(cm3)
Groups:
- Intensive Control of SBP: Participants randomized into the Intensive BP arm will have a goal of SBP <120 mm Hg. 2-drug therapy initiated in most Intensive participants; age ≥75 years and SBP 130-139 mm Hg on 0-1 drug; may begin with 1 drug, but add second at 1 month if SBP ≥130 mm Hg; drugs added and/or titrated at each visit (monthly) to achieve SBP <120 mm Hg; at periodic "milepost" visits: addition of another drug "required" if not at goal.
  Intensive control of SBP: Participants in the Intensive arm have a goal of SBP <120 mm Hg. Use of once-daily antihypertensive agents will be encouraged unless alternative frequency is indicated/necessary.
Arm/Group | Intensive Control of SBP | Standard Control of SBP
Number analyzed (Participants) | 200 | 249
asinh(cm3)
  Change in total white matter lesion volume from ba | 0.23 [0.17 to 0.29] | 0.37 [0.30 to 0.43]
  Change in total brain volume from baseline | -7.7 [-8.1 to -7.3] | -6.8 [-7.3 to -6.3]

ADVERSE EVENTS:
Time Frame: Includes Serious Adverse Events (SAEs) reported after randomization and throughout the duration of the trial, mean follow-up was 3.26 years.
Description: Adverse event reporting included occurrence of acute kidney injury or acute renal failure and specific monitored conditions if they were evaluated in emergency departments (hypotension, syncope, injurious falls, electrolyte abnormalities, bradycardia).
Arm/Group | Intensive Control of SBP | Standard Control of SBP
All-Cause Mortality (participants affected / at risk) | 155/4678 | 210/4683
Serious Adverse Events (participants affected / at risk) | 1793/4678 | 1736/4683
Other Adverse Events (participants affected / at risk) | 1399/4678 | 1342/4683
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive Control of SBP (N=4678) | Standard Control of SBP (N=4683)
Chest Pain (Cardiac disorders) | 198 | 191
Tachyarrhythmia (Cardiac disorders) | 141 | 176
Other ischaemic heart disease (Cardiac disorders) | 170 | 182
Death (General disorders) | 155 | 210
Knee arthroplasty (Musculoskeletal and connective tissue disorders) | 138 | 119
Ischaemic cerebrovascular conditions (Vascular disorders) | 109 | 121
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 100 | 114
Cardiac failure (Cardiac disorders) | 58 | 98
Myocardial infarcation (Cardiac disorders) | 70 | 106
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 42 | 64
Hip arthroplasty (Musculoskeletal and connective tissue disorders) | 67 | 81
Hypertension (Cardiac disorders) | 58 | 69
Urinary tract infection (Renal and urinary disorders) | 48 | 47
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 | 45
Dehydration (General disorders) | 51 | 41
Cellulitis (Infections and infestations) | 40 | 30
Sepsis (Infections and infestations) | 36 | 40
Spinal fusion surgery (Musculoskeletal and connective tissue disorders) | 46 | 30
Cardiac pacemaker insertion (Cardiac disorders) | 33 | 39
Spinal laminectomy (Musculoskeletal and connective tissue disorders) | 36 | 32
Pulmonary embolism (Vascular disorders) | 34 | 32
Dizziness (Nervous system disorders) | 34 | 25
Pulmonary embolism (Vascular disorders) | 32 | 31
Other (General disorders) | 952 | 951 — Occurred in less than 1% of total adverse events
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive Control of SBP (N=4678) | Standard Control of SBP (N=4683)
Hypotension (Cardiac disorders) | 48 | 27
Syncope (Nervous system disorders) | 56 | 33
Bradycardia (Vascular disorders) | 17 | 10
Electrolyte Abnormality (General disorders) | 33 | 22
Injurious fall (General disorders) | 229 | 222
Acute kidney injury or acute renal failure (Renal and urinary disorders) | 11 | 3
Serum sodium < 130 mmol/liter (General disorders) | 180 | 100
Serum sodium > 150 mmol/liter (General disorders) | 6 | 0
Serum potassium <3.0 mmol/liter (General disorders) | 114 | 74
Serum potassium >5.5 mmol/liter (General disorders) | 176 | 171
Orthostatic hypotension alone (Nervous system disorders) | 777 | 857
Orthostatic hypotension with dizziness (Nervous system disorders) | 62 | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-11-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT01206062/Prot_000.pdf
  • Informed Consent Form (2011-06-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT01206062/ICF_001.pdf